CLINICAL TRIAL: NCT01893476
Title: Tailored Implementation for Chronic Diseases.
Brief Title: A Pragmatic Cluster Trial of a Tailored Intervention to Improve COPD Management
Acronym: TICD-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, dr Maciej Godycki-Ćwirko, PhD, MD, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 258837
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; implementation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): In this arm, practitioners will provide usual care for COPD patients.
- adherence to guideline (Other): Implementation educational programme: guideline adherences. The results of this trial will be directly applicable to primary care settings. Should the interventions delivered at the level of the GP practice be found to be effective in improving patients' quality of life then the findings would have a wider application.
  Interventions: Other: Implementation educational programme

INTERVENTIONS:
Other: Implementation educational programme — Implementation educational programme will include: brief anti-smoking counseling, mMRC scale, checklist, training patient on correct use of inhaling. Participating physicians will receive training in brief anti-smoking counselling and will be asked to record information about. Additional form containing the mMRC dyspnoea scale will be inserted into patients' medical records. We will elaborate a checklist for practitioners with information about what should be done while consulting a patient with COPD. Investigators will provide practices with training inhaler and train staff. Practitioners will be asked to teach patients in correct use of each device. Practitioners will be asked to put this information to the patient's medical records.
  Other Names: implementation programme
  Arms: adherence to guideline

SUMMARY:
Background: Chronic Obstructive Pulmonary Disease (COPD) remains a major health problem, which is strongly related to smoking. Despite publication of guidelines on the prevention and treatment of COPD, not all COPD patients receive the best available healthcare. Investigators developed a tailored implementation strategy for improving primary care physicians' adherence to COPD management guidelines. The primary aim of the presented trial is to evaluate the effects of this strategy on physician's performance. The secondary aim is to examine the validity of the tailoring of implementation interventions.

Primary Trial Hypothesis: To study if the rate of adherence to the COPD guideline over a 1 year will increase among participants assigned to the intervention group in comparison to those assigned to the control group?

Methods/Design: A two-arm pragmatic cluster randomized trial is planned. A total of 540 patients with diagnosed COPD will be included from 18 general practices in Poland. A tailored implementation program will be offered to general practitioners. Participating physicians in the intervention practices (n=18) will receive training to provide brief anti-smoking counselling. An additional form containing COPD severity scale will be inserted into patient's medical records. The checklist with key information about the disease and its management while consulting a patient with COPD will be provided to practitioners. Investigators will provide practices with training inhaler devices for general practitioners (GPs) to teach patients in correct use of each device and to note this education/training in patient's medical records. The control practices will provide usual care.

Discussion: The results of this trial will be directly applicable to primary care in Poland and add to the growing body of evidence on interventions to improve chronic illness care.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) remains a major health problem. Worldwide it has been ranked as the sixth leading cause of death for both genders. In 2020 COPD is projected to rank fifth worldwide in burden of disease. It is also projected to be the fourth leading cause of death worldwide by 2030 due to an increase in smoking rates and demographic changes in many countries. The national survey conducted in Poland in 2007 indicated that 34% of men smoked daily, 2% were occasional smokers, 19% were former smokers and 45% never smoked. In women, these percentages were, respectively, 23%, 3%, 10% and 64%. Although COPD has received increasing attention from the medical community in some countries in recent years, it is still relatively unknown or ignored by the public as well as many healthcare providers and government officials.

Epidemiological studies of COPD on a representative sample have not been performed in Poland, but estimates from smaller suggested a relatively high prevalence. Studies which covered a selected geographical population found that signs and symptoms of COPD are seen in about 10% of patients over 40 years old. Studies in big cities in Poland showed a 9,8% prevalence of COPD in populations between 41 and 72 years old. These data are similar to European data, describing prevalence rates of 4-11% of COPD in adults in Europe. The absolute number of people suffering from COPD in Poland is estimated on about 2 million. This places COPD as the third most frequent - concerning frequency - chronic illness, and it is the fourth most common cause of death in Poland.

In Poland, many guidelines on COPD are used, some of which are national and some are international. There is no guideline in Poland which is designed for primary care.

Implementation of interventions directed on health professionals knowledge programme can change the professionals behavior. In this study the support strategy is applied to improve implementation process.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed COPD via the medical records with code J44

Exclusion Criteria:

* terminal illness
* cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The percentage of selected patients receiving anti-tabacco counseling recorded by the GPs in the labeled patients' medical records. | 1 year
  Brief anti-smoking counseling will be provided for GPs.

SECONDARY OUTCOMES:
Health outcomes in patients' medical records. | 1 year
  Investigators will review COPD patients' medical records to measure health outcomes such as smoking status change, quantity of and adherence to medication, change in modified Medical Research Council (mMRC) scale and number of exacerbations in the past and over the study period.
  Also, investigators will consider utilization of the Chronic Respiratory Questionnaire (CRQ).

OTHER OUTCOMES:
Adherence to the selected guidelines by GPs in primary care settings. | 1 year
  The percentage of GPs adhering to the selected guidelines in primary care settings.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Godycki-Cwirko, MD, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

REFERENCES:
- [Derived] Godycki-Cwirko M, Zakowska I, Kosiek K, Wensing M, Krawczyk J, Kowalczyk A. Evaluation of a tailored implementation strategy to improve the management of patients with chronic obstructive pulmonary disease in primary care: a study protocol of a cluster randomized trial. Trials. 2014 Apr 4;15:109. doi: 10.1186/1745-6215-15-109. PMID 24708623